CLINICAL TRIAL: NCT06017050
Title: Developing a Bullying Prevention Program That Transcends Physical Boundaries
Brief Title: BullyDown, a Text Messaging-based Bullying Prevention Program for Middle School-aged Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21HD104369 (NIH); R21HD104369 (NIH)
Record Dates: First submitted 2023-08-16; First posted 2023-08-30 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-07

CONDITIONS: Bullying
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Intervention Model Description: Youth will be randomized to either the intervention or control group.
Who Masked: Participant
Masking Description: Youth assigned to the control group will receive message written to seem as if it is intervention content (i.e., address bullying behaviors).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BullyDown intervention (Experimental)
  Interventions: Behavioral: BullyDown
- Healthy lifestyle control (Placebo Comparator)
  Interventions: Behavioral: Attention-matched control

INTERVENTIONS:
Behavioral: BullyDown — BullyDown is an 8 week, text messaging-based prevention program aimed to prevent bullying behaviors among middle school-aged youth. Message content is based upon the social-emotional learning model.
  Arms: BullyDown intervention
Behavioral: Attention-matched control — The attention-matched control will receive the messages for the same number of days as the intervention. Content will talk about 'healthy lifestyle' topics, such as fitness and healthy social media use.
  Arms: Healthy lifestyle control

SUMMARY:
Given the limited impact of existing school-based interventions and the time associated with implementing them during school time, more efficient and effective intervention methods are needed. Programs that can be delivered to middle school youth irrespective of whether they are attending school physically or virtually may be especially relevant as school boundaries become more fluid. BullyDown addresses this critical need by providing a scalable program that could be quickly and cost-effectively disseminated nationally.

ELIGIBILITY:
Participants will: be enrolled in one of our partner schools, be in middle school (i.e., 7th or 8th grade) or between the ages of 12-14 years of age, be English-speaking, own their own cell phone, intend to have the same cell phone number for at least 3 months (this may or may not apply, depending on the number of youth who meet this criterion), and provide informed written assent. Non-English speakers and youth who do not have the reading ability to complete the screener are not eligible. Youth recruited from schools will also be required to have parental permission.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Innovative Public Health Research, San Clemente, California
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BullyDown intervention | Healthy lifestyle control
Started | 71 | 67
Completed | 69 | 66
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BullyDown Intervention | Healthy Lifestyle Control | Total
Number analyzed (Participants) | 71 | 67 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 71 | 67 | 138
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Boys | 21 | 16 | 37
  Girls | 38 | 41 | 79
  Nonbinary youth | 4 | 6 | 10
  Declined to answer | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 50 | 104
  Not Hispanic or Latino | 17 | 14 | 31
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 41 | 41 | 82
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 13 | 11 | 24
Bullying perpetration [Count of Participants; unit: Participants] — Bullying is defined as engaging in at least one of 6 behaviors 3 or more times in the past 30 days. The behaviors include: 1) Hitting, kicking, pushing or shoving someone; 2) Making threatening or aggressive comments to someone; 3) Calling someone mean names; 4) Making fun of someone or teasing someone in a nasty way; 5) Leaving someone out or not letting someone into a group because you were mad at someone or were trying to make someone upset; and 6) Spreading rumors about someone, whether they were true or not.
  Participants | 9 | 11 | 20
Aggression perpetration [Count of Participants; unit: Participants] — Aggressive behavior is defined as engaging in at least one of 6 behaviors 1-2 times in the past 30 days. The behaviors include: 1) Hitting, kicking, pushing or shoving someone; 2) Making threatening or aggressive comments to someone; 3) Calling someone mean names; 4) Making fun of someone or teasing someone in a nasty way; 5) Leaving someone out or not letting someone into a group because you were mad at someone or were trying to make someone upset; and 6) Spreading rumors about someone, whether they were true or not.
  Participants | 24 | 22 | 46
Bystander behavior [Mean (Standard Deviation); unit: units on a scale] — Bystander intentions are measured using the 5-item University of Illinois Willingness to Intervene scale. Each of the items is measured on a 4-point Likert scale, resulting in a sum that ranges from 5 - 20. A higher score reflects a greater willingness to intervene.
  units on a scale | 14.7 (2.4) | 15.3 (2.7) | 15.0 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Recruitment Rate
Description: If at least 75% of eligible participants assent to participate, this will be supportive of a hypothesis of feasibility. Note that a youth could assent and not be randomized if they did not complete the baseline survey.
Time Frame: Recruitment period
Population: 474 youth were identified as eligible.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Number of Participants Recruited: Overall Number of Participants Recruited represent all participants who were determined to be eligible to be included in the study
Arm/Group | Overall Number of Participants Recruited
Number analyzed (Participants) | 474
Participants | 202

2. Primary Outcome: Acceptability of the Intervention
Description: Youth were asked: "How likely are you to recommend BullyDown to other people your age?" Answers were collected on a 5-point Likert scale. The response option ranged from 1-5, with higher values reflecting greater acceptability. An average score of 4 or higher was deemed supportive of program acceptability.
Time Frame: Intervention end, 9 weeks after program enrollment
Population: Youth who provided data at the program end survey were included in the analyses.
Measure: Mean (Standard Deviation); unit: Average score on a 5-point likert scale
Arm/Group | BullyDown intervention | Healthy lifestyle control
Number analyzed (Participants) | 59 | 56
Average score on a 5-point likert scale | 3.7 (1.1) | 3.6 (1.0)

3. Primary Outcome: Feasibility: Retention at 3-month Follow-up
Description: A retention rate of 80% or higher was deemed to be supportive of a hypothesis of feasibility
Time Frame: 21 weeks post-randomization, 3 months after the 9-week program ended
Measure: Count of Participants; unit: Participants
Arm/Group | BullyDown intervention | Healthy lifestyle control
Number analyzed (Participants) | 71 | 67
Participants | 48 | 49

4. Secondary Outcome: Feasibility: Retention Rate at Program End
Description: A retention rate of 80% or higher was deemed supportive of a hypothesis of feasibility.
Time Frame: 9 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | BullyDown intervention | Healthy lifestyle control
Number analyzed (Participants) | 71 | 67
Participants | 59 | 56

5. Other Pre Specified Outcome: Rates of Bullying Perpetration in the Intervention Versus Control Group
Description: Bullying behaviors towards other youth the same age 3 or more times in the past 30 days
Time Frame: Reported bullying perpetration behavior in the past 30 days at the end of the 9 week program
Population: Youth who provided data at the program end survey were included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | BullyDown intervention | Healthy lifestyle control
Number analyzed (Participants) | 59 | 56
Participants | 7 | 7

6. Other Pre Specified Outcome: Rates of Aggressive Behavior in the Intervention Versus Control Group
Description: Youth who report aggressive acts towards others 1-2 times in the past 30 days
Time Frame: Reported aggressive behavior in the past 30 days at the end of the 9 week program
Population: Youth who provided data at the program end survey were included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | BullyDown intervention | Healthy lifestyle control
Number analyzed (Participants) | 59 | 56
Participants | 15 | 14

7. Other Pre Specified Outcome: Scores of Bystanding Behavior in the Intervention Versus Control Group
Description: Bystander intentions are measured using the 5-item University of Illinois Willingness to Intervene scale. Each of the items is measured on a 4-point Likert scale, resulting in a sum that ranges from 5 - 20. A higher score reflects a greater willingness to intervene.
Time Frame: Responses provided at the program end survey, 9 weeks after they were randomized
Population: Youth who provided data at the program end survey were included in the analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BullyDown intervention | Healthy lifestyle control
Number analyzed (Participants) | 59 | 56
units on a scale | 14.7 (2.9) | 15.0 (3.1)

ADVERSE EVENTS:
Time Frame: Each participant was followed for 21 weeks
Arm/Group | BullyDown intervention | Healthy lifestyle control
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/67
Other Adverse Events (participants affected / at risk) | 0/71 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT06017050/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT06017050/ICF_000.pdf